CLINICAL TRIAL: NCT04800666
Title: Effect of Stellate Ganglion Block Combined With Facial Nerve Block on the Treatment of Idiopathic Facial Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Clinical Professor, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202103102
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Facial Palsy
Keywords: Peripheral Facial Palsy; Stellate Ganglion Block; Facial Nerve Block
MeSH Terms: interventions — mecobalamin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facial Nerve Block Group (Experimental): Facial Nerve Block and oral Mecobalamin Tablets
  Interventions: Procedure: Facial Nerve Block; Drug: Mecobalamin Tablets
- Stellate Ganglion Block Group (Experimental): Facial Nerve Block and Stellate Ganglion Block and oral Mecobalamin Tablets
  Interventions: Procedure: Stellate Ganglion Block; Procedure: Facial Nerve Block; Drug: Mecobalamin Tablets
- D Group (Experimental): Facial Nerve Block
  Interventions: Procedure: Facial Nerve Block
- C Group (Other): control
  Interventions: Drug: Mecobalamin Tablets

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Patients underwent a stellate-ganglion block at the anterolateral aspect of the C6 vertebra. After local analgesia (lidocaine 2%), a 22-gauge Quincke needle was placed in the anterolateral aspect of the C6 vertebral body. When the needle contacted the bone, it was drawn back 1 mm. 5 mL of 0·5% ropivacaine was subsequently injected next to the stellate ganglion to produce a sympathetic block.The effect of the stellate-ganglion block on the sympathetic nervous system was confirmed by the presence of Horner's syndrome (ie, facial anhydrosis, enophthalmos, ptosis, swelling of the lower eyelid, miosis, and blood-shot conjunctiva), and an increase in the temperature of the right hand of at least 2°F from baseline.
  Arms: Stellate Ganglion Block Group
Procedure: Facial Nerve Block — Operator touching the location of the mastoid, in the external auditory canal just below the front of the mastoid vertical needling.When touch the surface of the mastoid,adjust the needle across the front of the mastoid then slow needling about 1cm.The pin located below the stylomastoid foramen, and then injected drugs 5mL ( mecobalamin injection 1mg；lidocaine 60mg； dexamethasone 10mg )
  Arms: D Group; Facial Nerve Block Group; Stellate Ganglion Block Group
Drug: Mecobalamin Tablets — oral Mecobalamin Tablets tid-8
  Arms: C Group; Facial Nerve Block Group; Stellate Ganglion Block Group

SUMMARY:
Peripheral facial palsy is caused by damage to the facial nerve at any site of the peripheral branches after the facial nucleus.Stellate ganglion block is performed to treat peripheral facial palsy because it increases blood flow and promotes nerve regeneration.Facial Nerve Block worked with elimination of local inflammation of nerve and oppression. Facial nerve block is a treatment that inject drugs into the damaged nerve around to eliminate local inflammation and compression of the nerve.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed by clinical and neurological assessment as one-sided simple facial

* Age 18 to 75 years
* HBGS above Ⅳ
* the course of IFP not over 7 days.

Exclusion Criteria:

* Coagulation dysfunction
* plate plate plate shape, quantity or abnormal function
* mental system diseases
* Gillan-Bahrain syndrome
* cancer, mumps, shingles infection, jaw facial pus lymph nodeitis, encephalitis, -cerebral hemorrhage and other diseases
* local infection or systemic infectious disease at the puncture site
* can not accept to nerve block

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline House-Brackmann | Baseline ,change from baseline House-Brackmann at 3 days,6 days,9 days,14 days,one month,two month
  The House-Brackmann scale is a nerve grading system developed in 1985 by Los Angeles otolaryngologists Dr. John W. House and Dr. Derald E. Brackmann. It is used to characterize the severity of a facial paralysis patient's symptoms.
Change from Baseline Sunnybrook | Baseline,change from baseline Sunnybrook at 3 days,6 days,9 days,14 days, one month,two month
  Sunnybrook is a new facial nerve function of subjective assessment system.It is based on both static and dynamic aspects.

CONTACTS AND LOCATIONS:
Overall Officials: zhuan zhang, professor, Principal Investigator — The Affiliated Hospital of Yangzhou University
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China